CLINICAL TRIAL: NCT04634019
Title: Financially-Incentivized Knowledge Assessments to Improve Provider Compliance With Treatment Guidelines: A Randomized Controlled Trial
Brief Title: Financially-Incentives to Improve Provider Compliance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: World Bank (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IncentLearn
Record Dates: First submitted 2020-11-06; First posted 2020-11-18 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Compliant Behavior; Morbidity;Infant
Keywords: financial incentives; provider behavior; vignettes
MeSH Terms: conditions — Cooperative Behavior

STUDY DESIGN:
Intervention Model Description: This will be a two-arm parallel trial - control vs intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Providers in control facilities will not receive any additional training or knowledge assessments.
- Financial incentive arm (Experimental): Providers in treatment facilities will be visited once a quarter for a knowledge assessment using vignettes. Facilities performing well in this assessment will receive a quarterly bonus payment, which will be distributed among providers.
  Interventions: Behavioral: Financially incentivized knowledge assessments

INTERVENTIONS:
Behavioral: Financially incentivized knowledge assessments — We will conduct quarterly provider knowledge assessments at selected health facilities and will pay facilities a financial bonus if providers perform well on these tests. For the intervention, 12 clinical vignettes were created. These vignettes cover typical patient cases such as malaria, diarrhea and respiratory infections, and assess providers' ability to correctly diagnose and treat hypothetical questions. All medical staff members will be informed hat every 3 month there will be a knowledge assessment based on these vignettes and that the results will determine the total bonus payment made to the facility.
  Other Names: Provider knowledge assessments
  Arms: Financial incentive arm

SUMMARY:
The main objective of this study is to assess whether making health financing streams conditional on provider performance on knowledge assessment can increase provider compliance with under-5 case management guidelines.

DETAILED DESCRIPTION:
The main idea of the intervention is to conduct quarterly provider knowledge assessments at health facilities and to pay facilities a bonus if providers perform well on these tests. For the intervention, 12 clinical vignettes were created. These vignettes cover typical patient cases such as malaria, diarrhea and respiratory infections, and assess providers' ability to correctly diagnose and treat hypothetical questions. All medical staff members were informed hat every 3 month there would be a knowledge assessment based on these vignettes and that the results would determine the total bonus payment made to the facility.

Each quarter, facilities receive a supervision visit. During the supervision visits, one provider is randomly chosen for the knowledge assessments, and is tested on two randomly chosen vignette cases.

In order to create a quarterly performance score, the scores on the two vignettes are then averaged. Fifty percent of the overall facility quality score is determined by the general quality checklist that captures basic structural and process features of the facility. The remaining fifty percent are directly determined by the providers' performance on the knowledge assessments. If the overall quality score is below 50%, no quality payments are made. If the quality score is >=50%, facilities can receive a top-up payment of up to 25% of the quantity-based payments. The total bonus percentage is determined by multiplying the quality score (with ranges between 0 and 100%) with the maximum 25% bonus.

ELIGIBILITY:
Inclusion Criteria:

* all providers working at the 110 facilities selected for the study will be included in the study.

Exclusion Criteria:

* none.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Compliance with integrated management of childhood illness (IMCI) guidelines | Endline (30 months after project start)
  Compliance will be measured through up to 8 direct observations of under-5 sick child visits at each facility collected over a four-day period. During each visit, trained observes will document how many of the 10 diagnostic steps specified in the WHO's Integrated Management of Child Illness (IMCI) are followed by the provider. Compliance will be defined as least 8 out of 10 diagnostic processes completed.

SECONDARY OUTCOMES:
Knowledge regarding IMCI guidelines | Endline (30 months after project start)
  Knowledge of IMCI guidelines will be assessed through vignettes administered to providers at baseline and endline. A total of five vignettes will be given to providers, each describing a scenario involving a sick child under age 5. An overall knowledge score will be created to measure the extent to which the diagnosis and treatment chosen by providers matches those specified in the nationally used Integrated Management of Child Illness guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Gil Shapira, PhD, Principal Investigator — World Bank
Locations (2):
- Congo Ministry of Public Health, Kinshasa, Democratic Republic of the Congo
- Swiss Tropical and Public Health Institute, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The data collected as part of this project will be made available to researchers through the World Bank's data repository.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Upon completion of study
Access Criteria: public access

REFERENCES:
- [Derived] Fink G, Fritsche G, Samaha H, Sese C, Shapira G. Financially incentivized knowledge assessments to improve provider compliance with treatment guidelines: a cluster-randomized controlled trial. Trials. 2022 Mar 21;23(1):227. doi: 10.1186/s13063-022-06129-8. PMID 35313932